CLINICAL TRIAL: NCT06271772
Title: Rose Bengal Electromagnetic Activation With Green Light for Infection Reduction II
Acronym: REAGIR II
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Stanford University (Other); Aravind Eye Care System (Other); Federal University of São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-26045-RII
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Bacterial Keratitis
MeSH Terms: interventions — Rose Bengal; Corneal Cross-Linking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RB-PDT Plus Early Steroids (Experimental)
  Interventions: Drug: Difluprednate Ophthalmic; Drug: Rose Bengal; Drug: Moxifloxacin Ophthalmic
- Sham RB-PDT Plus Early Steroids (Experimental)
  Interventions: Drug: Difluprednate Ophthalmic; Drug: Moxifloxacin Ophthalmic

INTERVENTIONS:
Drug: Difluprednate Ophthalmic — Difluprednate 0.05% is a corticosteroid used to reduce inflammation in the eye. Participants will receive one drop of 0.05% difluprednate four times daily beginning 24 hours after the initiation of antibiotics for 1 week, decreased by 1 drop weekly for a total of 4 weeks of steroid therapy.
Drug: Rose Bengal — Study participants receive RB-PDT within 48 hours of randomization. All participants will receive a 30-minute loading dose of topical Rose Bengal (0.1% RB in 0.9% sodium chloride) which will be applied in 3-minute intervals to the de-epithelialized cornea. This will be followed by irradiation with a 6mW/cm2 custom-made green LED source for 15 minutes (5.4J/cm2). Repeat cornea culture will be collected within 24 hours after the procedure.
  Other Names: Corneal Cross Linking with rose Bengal
  Arms: RB-PDT Plus Early Steroids
Drug: Moxifloxacin Ophthalmic — Topical moxifloxacin 0.5% is a fluoroquinolone antibiotic that is used to treat bacterial infections. This is a standard therapy for bacterial keratitis.

SUMMARY:
Rose Bengal Electromagnetic Activation with Green light for Infection Reduction II (REAGIR II) is a randomized, double-masked feasibility study. The purpose of this study is to determine differences in 6-month visual acuity between medical antimicrobial treatments alone versus antimicrobial treatment plus cross-linking with rose Bengal (RB-PDT).

Patients presenting to one of the Aravind Eye Hospitals in India or to the Federal University of São Paulo ophthalmology clinic in Brazil with smear-positive and/or culture positive typical (I.e. non-Nocardia or Mycobacteria) bacterial corneal ulcers and moderate to severe vision loss, defined as Snellen visual acuity of 20/40 of worse, will be eligible for inclusion. Those who agree to participate will be randomized to one of two treatment groups:

* Group 6, RB-PDT Plus Early Steroids: topical 0.5% moxifloxacin plus topical difluprednate 0.05% plus RB-PDT
* Group 7, Sham RB-PDT Plus Early Steroids: topical 0.5% moxifloxacin plus topical difluprednate 0.05% plus sham RB-PDT

ELIGIBILITY:
Inclusion Criteria:

* Corneal ulcer that is smear positive and/or culture positive (within 24 hours) for typical bacteria (i.e. non-Nocardia or Myobacteria)
* Moderate to severe vision loss, defined as Snellen visual acuity of 20/40 (6/12) or worse
* Corneal thickness ≥350 µm, as measured on AS-OCT
* Age over 18 years
* Basic understanding of the study as determined by the physician
* Commitment to return for follow up visits

Exclusion Criteria:

* Evidence of concomitant infection on exam, gram stain, or confocal microscopy (i.e. herpes, both bacteria and acanthamoeba on gram stain)
* Impending or frank perforation at recruitment
* Involvement of sclera at presentation
* Presence of desmetocele at recruitment
* Non-infectious or autoimmune keratitis
* History of corneal transplantation
* History of intraocular surgery within the last three months*
* Pinhole visual acuity worse than 20/200 in the unaffected eye
* Participants who are decisionally and/or cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Best Spectacle-Corrected Visual Acuity | 6 months
  Best Spectacle-Corrected Visual Acuity

SECONDARY OUTCOMES:
Best Spectacle-Corrected Visual Acuity | 3 Weeks, 3 Months, 12 Months
  Best Spectacle-Corrected Visual Acuity
Scar size | 3 Weeks, 3 Months, 6 Months 12 Months
  Geometric mean
Scar depth | 3 Weeks, 3 Months, 6 Months 12 Months
  Geometric mean
Adverse Events | 12 Months
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rose-Nussbaumer, MD, Principal Investigator — Stanford University; Thomas Lietman, MD, Principal Investigator — University of California, San Francisco; Nicole Varnado, MPH, Study Director — Stanford University
Locations (2):
- Federal University of São Paulo, São Paulo, Brazil
- Aravind Eye Care System, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No